CLINICAL TRIAL: NCT06546462
Title: Can a Specific OMT Protocol Influence Patient-reported Pain and Associated Analgesia Use for Primary Headache Disorders?
Brief Title: Can a Specific OMT Protocol Influence Patient Pain and Associated Analgesia Use for Primary Headache Disorders?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Headache OMT; BHS-1852 (Other: New York Institute of Technology BHS-IRB)
Record Dates: First submitted 2023-11-13; First posted 2024-08-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Headache Disorders; Headache; Analgesia; Opioid Use; Osteopathy
Keywords: Osteopathic manipulative medicine; Osteopathic manipulative treatment; Headache
MeSH Terms: conditions — Headache Disorders; Headache; Agnosia | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulation arm (Experimental): * All subjects receive osteopathic structural exam and screening for somatic dysfunction of the cranium, spine, sacrum, and ribs.
  * The OMT arm will have the following techniques performed for the stated time to total 14 minutes.
    1. Thoracic inlet release: 45 seconds maximum
    2. Suboccipital release: 1 minute maximum
    3. Occipito-mastoid suture release: 1 minute maximum
    4. Venous sinus drainage: 1 minute maximum
    5. Balanced membranous tension: 1 minute maximum
    6. Compression of the 4th Ventricle (CV4): 1 minute maximum
    7. Cervical soft tissue: 1 minute maximum
    8. Trapezius inhibition: 45 seconds maximum
    9. Bilateral rib raising: 2 minutes max (1 min per side)
    10. Sacroiliac gapping: 1 minute maximum
    11. Sacral rock: 1 minute maximum
    12. Seated bilateral thoracic and lumbar paraspinal articulation: 2 minutes maximum
  Interventions: Other: Osteopathic Manipulative Treatment (OMT)
- Sham Light touch arm (Sham Comparator): * All subjects receive osteopathic structural exam and screening for somatic dysfunction of the cranium, spine, sacrum, and ribs..
  * The sham group will follow an established protocol of light systematic touch for the same duration as the OMT group. It consists of contacting a sequence of anatomical areas for 2 minutes each: right ankle, left knee, right hip, diaphragm, right shoulder, neck, and cranium. Total procedure time is 14 minutes.
  Interventions: Other: Sham Light touch arm

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment (OMT) — The active arm will receive osteopathic manipulative treatment which is a hands-on treatment modality use to treat a variety of health concerns.
  Arms: Osteopathic Manipulation arm
Other: Sham Light touch arm — Sham arm will receive a light touch sham treatment.
  Arms: Sham Light touch arm

SUMMARY:
The purpose of this study is to see if osteopathic manipulation or light touch can reduce either or both frequency of headaches or use of pain medication. Osteopathic manipulative treatment (OMT) has been shown to help headache symptoms. The investigators like to see if regular OMT sessions can help reduce headache discomfort and also reduce use of pain medication like over-the-counter medications, migraine medications, and opioids. In this randomized controlled trial, a set sequence of OMT will be compared to light touch sham protocol. Investigators will compare participant responses to questionnaires that assess items including pain levels and reported pain medication use for the course of the study period to see if there are any shifts.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of osteopathic manipulative treatment protocol (OMT) or light touch protocol in reducing headache frequency and the use of pain medication for headache pain. Previous research has suggested that OMT may alleviate headache symptoms. This randomized controlled trial aims to determine whether regular OMT sessions can decrease headache discomfort and reduce the use of pain medications, including over-the-counter medications, migraine-specific treatments, and opioids. The study consists of a ten-week period, including 2 weeks of observation, 6 weeks of intervention, and 2 weeks of washout. Participants will be randomly assigned to either receive OMT or a light touch protocol. Investigators will compare questionnaires assessing quality of life and functionality scales. Pain levels and medication use will be logged daily throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* takes opioids or any other pain medication for headaches more than 10 times a month (including over the counter and prescription medications for headaches).
* 3 months or greater history of headaches or migraines
* Patient able to tolerate OMT based on osteopathic physician discretion and with consideration of absolute and relative contraindications to OMT

Exclusion Criteria:

* current diagnosis of neoplasm
* history of headache secondary to trauma or concussion
* history of brain/cranial surgery, cerebral vascular events/disease (e.g., stroke, Brain arteriovenous malformation (AVM), vertebral artery disease)
* acute psychiatric diagnosis
* pregnancy
* history of substance use disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain levels | Assessment of weekly average pain from week 1 till week 10 end of the study period
  The primary outcome measures will assess if consistent use of OMT for headache causes a reduction in headache pain for headache-associated discomfort. Pain will be rated on a Numeric Rating Scale (NRS) so individuals can rate their pain on a scale from 0 (no pain) to 10 (worst possible pain).
Change in analgesia use | Assessment of weekly amount of pain medications used from week 1 till week 10 end of the study period
  The primary outcome measures will assess if consistent use of OMT for headache causes a reduction in headache analgesia use for headache-associated discomfort.

SECONDARY OUTCOMES:
Change in quality of Life - Headache disability index | To be completed at Week 1 (initial visit), week 6 (midpoint of study), and week 10 (at completion of study)
  Secondary measures will assess any changes to physical and mental health and reduce the impact of headaches via the Headache disability index. Max score = 100. The higher the score the worse the symptoms. A 29 point change (95% confidence interval) or greater in the total score from test to retest must occur before the change can be attributed to treatment effects.
Change in quality of Life - Headache Impact Test (HIT-6) | To be completed at Week 1 (initial visit), week 6 (midpoint of study), and week 10 (at completion of study)
  Secondary measures will assess any changes to physical and mental health and reduce the impact of headaches via the Headache Impact Test (HIT-6) Higher scores indicate a greater impact on your life. Score range 36-78.
Change in quality of Life - The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group (EQ-5DL) | To be completed at Week 1 (initial visit), week 6 (midpoint of study), and week 10 (at completion of study)
  Secondary measures will assess any changes to physical and mental health and reduce the impact of headaches via EQ-5DL - quality of life measure. 5 questions rated on levels with 5 being the highest level of disability and an additional questions on overall health rated on a scale of 100 with 100 being the best possible health and 0 being being the worst possible health.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Yao, D.O, Principal Investigator — New York Institute of Technology
Locations (1):
- Riland Academic Health Care Center, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jara Silva CE, Joseph AM, Khatib M, Knafo J, Karas M, Krupa K, Rivera B, Macia A, Madhu B, McMillan M, Burtch J, Quinonez J, Albert T, Khanna D. Osteopathic Manipulative Treatment and the Management of Headaches: A Scoping Review. Cureus. 2022 Aug 9;14(8):e27830. doi: 10.7759/cureus.27830. eCollection 2022 Aug. PMID 36110479
- [Background] Chin J, Qiu W, Lomiguen CM, Volokitin M. Osteopathic Manipulative Treatment in Tension Headaches. Cureus. 2020 Dec 12;12(12):e12040. doi: 10.7759/cureus.12040. PMID 33457139